CLINICAL TRIAL: NCT01120730
Title: Fluid Resuscitation With HES 200/0.5 10% in Severe Burn Injury
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Thomas A. Neff, Surgical ICU University Hospital Zurich
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: USZ-BURN; 97/x (Other: kantonale Ethikkommision)
Record Dates: First submitted 2010-04-28; First posted 2010-05-11 (Estimated); Last update posted 2010-05-11 (Estimated); Status verified 2010-05

CONDITIONS: Survival; Renal Failure
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HES (Active Comparator): Fluid resuscitation with HES
  Interventions: Drug: fluid resuscitation
- ringers lactat (Placebo Comparator): Standard treatment
  Interventions: Drug: Fluid resuscitation

INTERVENTIONS:
Drug: fluid resuscitation — fluid resuscitation with HES
  Arms: HES
Drug: Fluid resuscitation — Fluid resuscitation in standardized fashion
  Arms: ringers lactat

SUMMARY:
HES 200/0.5 10% is equal to ringers lactat solution.

DETAILED DESCRIPTION:
30 Patients were enrolled to the study, either to the hyperoncotic HES 200/0.5 (10%) group or to the crystalloids only group. After a treatment protocol of 72 hours we collected data about complications like pulmonary failure and abdominal compartment syndrome. Furthermore, we addressed the question of incidence of mortality and renal failure.

ELIGIBILITY:
Inclusion Criteria:

* All burn victims with burned surface area bigger than 20%

Exclusion Criteria:

* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 1997-04; Primary Completion 1998-09 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Intensive care unit mortality | 28 days
  28 days

SECONDARY OUTCOMES:
fluid amount during the first 72 hours | 28 days
  Fluid resuscitation after burn

CONTACTS AND LOCATIONS:
Overall Officials: Markus Béchir, md, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Bechir M, Puhan MA, Neff SB, Guggenheim M, Wedler V, Stover JF, Stocker R, Neff TA. Early fluid resuscitation with hyperoncotic hydroxyethyl starch 200/0.5 (10%) in severe burn injury. Crit Care. 2010;14(3):R123. doi: 10.1186/cc9086. Epub 2010 Jun 28. PMID 20584291